CLINICAL TRIAL: NCT02462499
Title: Eplerenone Treatment for Chronic Central Serous Chorioretinopathy in Hungarian Population
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Semmelweis University (Other)
Responsible Party: Principal Investigator, Dr. Ecsedy, Assistant Professor, Semmelweis University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSCR 104/2014
Record Dates: First submitted 2015-05-26; First posted 2015-06-04 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Chronic Central Serous Chorioretinopathy
MeSH Terms: interventions — Eplerenone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Treatment: Eplerenone (Inspra) All patients will receive 25mg eplerenone once a day for a week, followed by 50mg once a day, for a total of 4-12 weeks.
  Interventions: Drug: Inspra (eplerenone)

INTERVENTIONS:
Drug: Inspra (eplerenone)

SUMMARY:
The aim of the study is to determine the efficacy and safety of treatment with the drug eplerenone in patients with chronic central serous chorioretinopathy.

ELIGIBILITY:
Inclusion Criteria:

* Chronic central serous chorioretinopathy (CSCR) with persistent subretinal fluid on OCT for more than 3 months after initial presentation .
* Written informed consent

Exclusion Criteria:

* Persons with impaired decision-making ability.
* Pregnant women or who are actively trying to conceive.
* Additional eye disease affecting the macula or posterior retina.
* Creatinine clearance < 50 ml/min
* Hyperkalemia > 5 mmol/l
* Serum creatinine > 2 mg/dl in men or > 1.8 mg/dl in women
* Treatment with potassium sparing agents or potassium
* Treatment with any other drugs known to cause interaction with eplerenone
* Microalbuminuria in patients with type 2 diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2014-06; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Resolution of sub-retinal fluid measured by optical coherence tomography (OCT). | 6 months
Number of Participants with Adverse Events as a Measure of Safety and Tolerability. | 3 months

SECONDARY OUTCOMES:
Changes in macular volume at baseline, during and after the treatment with eplerenone. | 6 months
Changes in visual acuity at baseline measured on Early Treatment of Diabetic Retinopathy Study (ETDRS) chart, during and after the treatment with eplerenone. | 6 months
Changes in choroideal thickness at baseline measured by OCT, during and after the treatment with eplerenone in both eyes. | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Semmelweis University, Department of Ophthalmology, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No